CLINICAL TRIAL: NCT03052179
Title: The Clinical and Biological Effects Of The Use Of Probiotic VSL#3 In Patients With Oral Lichen Planus : a Proof-of-concept Study
Brief Title: The Clinical and Biological Effects Of The Use Of Probiotic VSL#3 In Patients With Oral Lichen Planus
Acronym: CABRIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16/0622
Record Dates: First submitted 2017-02-09; First posted 2017-02-14 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, placebo-controlled
Who Masked: Participant, Investigator
Masking Description: Either participant or the investigator will be blinded. The key of randomisation will be held by the third statistician party, and the company which supply and labeled the product study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VSL#3 (Active Comparator): VSL#3 poly-biotic 450 billion in sachet orally, two sachets in the morning and two sahcets in the evening for 30 days
  Interventions: Dietary Supplement: Poly-biotic
- Placebo (Placebo Comparator): Maltose in sachet orally, two sachets in the morning and two sahcets in the evening for 30 days
  Interventions: Dietary Supplement: Poly-biotic

INTERVENTIONS:
Dietary Supplement: Poly-biotic — Before-after treatment
  Other Names: VSL#3 5015919450087

SUMMARY:
Oral Lichen Planus (OLP) is an inflammatory disease of mucosal and skin with unknown etiology. The prevalence rate in England is reported to be between 1-2.4%. OLP contributed to around 40% of all visits or 1,200 appointments in 2014 at the Eastman Dental Hospital. Pain, discomfort, long-standing use of medications, lesion recurrence and adverse side effects of therapy are commonly associated with OLP, eventually leading to a significant reduction in a patient quality of life. In addition, there is also increased risk of developing oral cancer in patients with OLP. The current gold standard treatment for OLP is corticosteroid, which can result in adverse side effects including increased risk of infections and skin cancer, reduced systemic immune system, and hepatotoxicity with long-term usage.

Alternatively, a probiotic food supplement, VSL#3, has shown evidence of been able to induce and maintain remission in Inflammatory Bowel Disease (IBD), with no adverse effect a part than bloating, reported. Additionally, a preliminary report shown that probiotics treatment in Behcet's disease and Recurrent Aphthous Stomatitis (RAS) lesion resulted in reducing the number of oral ulcerations and subjective relief of oral discomfort.

Investigator designed a clinical trial with 30 participants allocated to one of two interventions, VSL#3 or placebo. Individuals with biopsy-confirmed OLP who experience painful symptoms will be recruited from a single site research site (Eastman Dental Hospital (EDH)). Either the active VSL#3 or the placebo, provided by Ferring Pharmaceuticals Limited, will be consume twice a day over a 30 days period. Questionnaires that will determine pain levels, disease activity and quality of life will be completed before the study begins, on days 15, 30 and 30 days after the last supplement intake. In addition saliva and blood samples will be taken before therapy begin, at 30 days of therapy, and 30 days after the last supplement intake. The levels of pro-inflammatory cytokines and the oral microbiota will be investigated using these samples. A blinded clinician will assess the clinical effects between groups of active VSL #3 and placebo and the results will analyze by statistician.

DETAILED DESCRIPTION:
Primary objective:

• To investigate the effects of 30 days use of supplement therapy of probiotic VSL#3 on painful symptoms of OLP at the end of the therapy (30-days endpoint) and 30 days after the last dose (60-days endpoint).

Secondary objective:

1. To investigate the effects of 30 days use of supplement therapy of probiotic VSL#3 on OLP disease activity.
2. To investigate the effect of 30 days use of supplement therapy of probiotic VSL#3 on quality of life.
3. To investigate acceptability of the intervention and potential adverse effects. and for the mechanistic study, whether :

   * The use of VSL#3 is associated with metagenomics changes in saliva.
   * The use of VSL#3 is associated with changes in the serum expression profile of pro-inflammatory cytokines.

A randomized, double blinded, placebo-controlled trial study on individuals with OLP.

Patients with painful ulcerative biopsy-confirmed OLP attending the Oral Medicine clinics of the UCLH ( University college of London hospital) Eastman Hospital and meeting the inclusion criteria of the study will be given information about the trial and invited to participate.

30 individuals who consent will be recruited and randomised in two groups: group A (15 participants) will receive the VSL#3 and group B (15 participants) will receive a placebo. A centralised computer-generated randomization list provided by an independent third party will be used to conceal allocation of patients to the treatments. The list will be sent to the drug manufacturer who will label the VSL#3 or placebo with relevant study participant code, which will come in the same identical plain-packages to ensure blinding (neither the participants nor the investigator will be aware of the sachets content). The study statistician will also be blinded to the allocation. Patients will be allowed to use best standard therapy during the study.

To demonstrate the research hypotheses, Investigators will record oral painful symptoms, disease activity, and quality of life in participants before, at 15 and 30 days from treatment start, and 30 days (day 60) after the last VSL#3 supplement intake.

60 days + 15 days 21 months Single-site 30 participants

Inclusion Criteria:

1. Biopsy-proven diagnosis of OLP as per WHO histological criteria* with no evidence of epithelial dysplasia or malignancy.
2. Presence of painful oral symptoms associated to OLP, with minimum severity of pain being 3 or more, on a 0-10 numeric pain rating scale at screening and confirmed at recruitment/start of the intervention.
3. Age >18 years and willing to participate into the study.
4. Receiving no therapy or receiving best standard topical therapy (typically topical corticosteroids or immunosuppressant) with the exclusion of systemic corticosteroids or systemic immunosuppressant.

   * I. R. H. Kramer, R. B. Lucas, J. J. Pindborg, and L. H. Sobin, "Definition of leukoplakia and related lesions: an aid to studies on oral precancer," Oral Surgery Oral Medicine and Oral Pathology, vol. 46, no. 4, pp. 518-539, 1978

Exclusion Criteria

1. The use of systemic antibiotics, retinoid, corticosteroids or immunosuppressant within four weeks prior to enrolment in the study.
2. Pregnancy* or receiving IVF treatment.
3. Individuals with known history of systemic disorders affecting the immune system (e.g., connective tissue disorders, cancer, etc.)
4. Active cancer or cancer in remission undergoing maintenance with chemotherapy or immunomodulatory agents.
5. Evidence of oral epithelial dysplasia or malignancy on previous biopsy.

   * Evidence of negative pregnancy test at screening / randomization visit (strip urine test) in women of child-bearing age in which the possibility of being pregnant cannot be otherwise excluded.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven diagnosis of OLP as per WHO histological criteria* with no evidence of epithelial dysplasia or malignancy.
2. Presence of painful oral symptoms associated to OLP, with minimum severity of pain being 3 or more, on a 0-10 numeric pain rating scale at screening and confirmed at recruitment/start of the intervention.
3. Age >18 years and willing to participate into the study.
4. Receiving no therapy or receiving best standard topical therapy (typically topical corticosteroids or immunosuppressant) with the exclusion of systemic corticosteroids or systemic immunosuppressant

Exclusion Criteria:

1. Use of systemic antibiotics, retinoid, corticosteroids or immunosuppressant.
2. Pregnancy or receiving IVF treatment.
3. Individuals with systemic disorders affecting the immune system (e.g., HIV, connective tissue disorders, cancer, etc.)
4. Evidence of oral dysplasia or malignancy on previous biopsy. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
pain - Numeric Rating Scale (NRS) | 30 days
  is a 10 point scale for participant self-reporting pain. Participant will asked to point out the scale from 0 = no pain and 10 = worse pain can imagine.

SECONDARY OUTCOMES:
ESS | 30 days
  Escudier's scoring system to measure disease activity based on size and number of lesion
COMDQ | 30 days
  Validated questioner for chronic oral mucosal disease

OTHER OUTCOMES:
Metagenomic changing in saliva | 30 days
  To observed changing of bacterial composition before and after treatment
Cytokine serum level | 30 days
  To observed changing in serum level cytokine before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Smith, Dr, Principal Investigator — University College, London
Locations (1):
- University College of London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
the data will be kept anynomous. This data only accessible by the party mention in the protocols